CLINICAL TRIAL: NCT06502665
Title: Outcomes From Secondary Ovulation Induction Following Failed Oocyte Pick-up IVF Cycles
Brief Title: Second Ovulation Induction
Status: Completed | Type: Observational
Sponsor: Clinique Ovo (Industry)
Responsible Party: Sponsor
Other Study IDs: 3572
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2024-07

CONDITIONS: IVF; Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Women having had second ovulation induction after failed oocyte pick-up — IVF success is defined by the number of retrieved oocytes. Identifying women at risk of failed oocyte pick-up at the first oocyte pick-up and optimizing their ovulation induction could enhance outcomes

SUMMARY:
Studies reported various risk factors for inadequate ovulation induction such as body mass index, low ovarian reserve, low baseline FSH and LH, and previous use of contraception or agonist.

The flexibility to use human chorionic gonadotropin (hCG) or gonadotropin-releasing hormone agonist (GnRHa) in ovulation induction for antagonist protocol or progestin primed ovarian stimulation (PPOS) is an advantage helping fertility doctors to decrease the risk of ovarian hyperstimulation syndrome. However, luteinizing hormone (LH) levels <15UI/L and progesterone ≤11.13nmol/L eight to twelve hours post GnRHa trigger were highly correlated to failed oocyte pickup (FOP).

Rescue hCG have been found to increase favorable outcomes in patients with FOP. The presence of false FOP could be due pharmaceutical reasons and human error. Genuine FOP could be due to intrinsic ovarian pathology.

The FOP is defined as the absence of oocytes after ovarian stimulation and follicular aspiration. It is an uncomfortable situation for the patient and medical team to deal with due to the apparent expectations of favorable results.

Ovulation induction could be via GnRHa, HCG, or both in antagonist protocol and PPOS protocol. Long or short agonist protocol could be triggered only via HCG.

ELIGIBILITY:
Inclusion Criteria:

* Participants with no oocytes retrieved in the first ovum pick-up

Exclusion Criteria:

* Error in trigger medication or timing by the patient/ medical team
* Major absence of information (primary objective, trigger medication, time interval of trigger and ovum pick-up

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Women able to have oocyte retrieval after in-vitro fertilization
Study Population: Electronic medical record from 2018 to 2023 of patients having undergone an IVF cycle
Sampling Method: Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2024-07-04 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Oocyte pick-up at retrieval | 36 hours after ovulation triggering
  Number of retrieved oocytes after second ovulation induction in patients with FOP

SECONDARY OUTCOMES:
Timing of ovulation triggering | 24 to 36 hours after ovulation triggering
  Time interval outcomes between trigger and ovum pickup

CONTACTS AND LOCATIONS:
Overall Officials: Simon Phillips, PhD, Principal Investigator — Clinique Ovo
Locations (1):
- Clinique Ovo, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No